CLINICAL TRIAL: NCT04470063
Title: A Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multi-dose DDO-3055 Tablets in Patients With Anemia of Non-dialysis Chronic Kidney Diseases-Randomized, Double-blind, Dose Escalation, Placebo Controlled Phase I Clinical Trial.
Brief Title: Multi-dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DDO-3055 Tablets in Patients With Anemia of Non-dialysis Chronic Kidney Diseases.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DDO-3055-104
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Anemia Associated Chronic Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental)
  Interventions: Drug: DDO-3055 tablets; Drug: Placebo
- group B (Experimental)
  Interventions: Drug: DDO-3055 tablets; Drug: Placebo
- group C (Experimental)
  Interventions: Drug: DDO-3055 tablets; Drug: Placebo

INTERVENTIONS:
Drug: DDO-3055 tablets — Multi-dose for DDO-3055 tablets
Drug: Placebo — Multi-dose for Placebo

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multi-dose DDO-3055 tablets in patients with anemia of non-dialysis chronic kidney diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD anemia aged 18-70 years who were not on dialysis and were not expected to undergo dialysis during the study period, regardless of gender;
* Male weight≥50kg, female weight≥45kg, and 19kg/m2≤BMI<28kg/m2;
* Signed informed consent.

Exclusion Criteria:

* Allergic constitution, suspected to be allergic to the study drug or any component in the study drug;
* Patients with acute coronary syndrome, stroke, thromboembolism (such as deep vein thrombosis or pulmonary embolism) or a history of seizures within 6 months before screening;
* Patients with uncontroll ed hypertension;
* New York Heart Association grade III or IV congestive heart failure at the time of screening;
* ALT,AST or total bilirubin exceeds 1.5 times the upper limit of normal value (ULN) during the screening period;
* Suffer from anemia other than CKD.
* Patients with a history of chronic liver disease;
* Patients with active bleeding or known coagulopathy;
* Patients who have any previous organ transplant or plan to perform organ transplant;
* Intravenous iron supplementation within 1 month before screening;
* Used erythropoiesis stimulator (ESAs), hypoxia-inducible factor-prolyl hydroxylase inhibitor (HIF-PHI), androgen, blood transfusion therapy within 3 months before screening;
* Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, and human immunodeficiency virus (HIV) antibody were positive;
* Patients with blood loss ≥400mL within 3 months before screening;
* Subjects who have taken other clinical trial drugs or are expected to have a legacy effect of the trial treatment;
* Participants who are unwilling to take contraception or male subjects who cannot guarantee not to donate sperm during the trial and within 30 days after the last dose; female subjects with fertility who did not use contraception for at least 14 days before dosing;or male and female subjects who did not agree to use physical contraception during the trial;
* Patients who had a positive blood pregnancy test and were breastfeeding at the time of screening;
* According to the study physician's judgment, there may be any other anemia factors that may exist, any possibility to increase the risk of the study, affect the subject's compliance with the protocol, or affect the physical or psychological disease or condition of the subject to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events to assess safety and tolerability. | up to 37 days

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat Sen memorial hospital Sun Yat Sen university, Guangzhou, Guangdong
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Henbei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Zhongda Hospital Southeast Universtiy, Nanjing, Jiangsu
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shandong Qianfo Mountain hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan